CLINICAL TRIAL: NCT07223086
Title: Use of Tinted Contact Lenses for Concussion-Related Light Sensitivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Candice Turner, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015049; Faculty development grant (Other Grant/Funding Number: Faculty development grant)
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Concussion, Mild; Photophobia; Contact Lens
Keywords: Mild concussion; tinted contact lenses; light sensitivity
MeSH Terms: conditions — Brain Concussion; Photophobia | interventions — Contact Lenses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participants with concussion and light sensitivity fit with broad band (clear) contact lens (Active Comparator): UPSIS-2 scale 15-60, eligible participants score greater than or equal to 26 are fit in broad band (clear) contact lenses.
  Interventions: Device: broad band (clear) contact lenses
- Participants with concussion and light sensitivity fit with narrow band (tinted) contact lens (Active Comparator): UPSIS-2 scale 15-60, eligible participants score greater than or equal to 26 are fit in narrow wavelength (tinted) contact lenses.
  Interventions: Device: Narrow band (tinted) contact lenses

INTERVENTIONS:
Device: Narrow band (tinted) contact lenses — Participants will receive these contacts based on the results of the Utah Photophobia Symptom Impact Scale (survey).
  Other Names: Altius contact lenses
  Arms: Participants with concussion and light sensitivity fit with narrow band (tinted) contact lens
Device: broad band (clear) contact lenses — Participants will receive these contacts based on the results of the Utah Photophobia Symptom Impact Scale (survey).
  Other Names: BioTrue One Day; Infuse daily disposable contact lenses; Clariti 1 Day clear contact lenses
  Arms: Participants with concussion and light sensitivity fit with broad band (clear) contact lens

SUMMARY:
The purpose of this study is to gather pilot data on the effectiveness of daily disposable tinted contact lenses in reducing photophobia (light sensitivity) following a concussion, with the goal of facilitating the return to work or school.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed mild traumatic brain injury (concussion)
* age 18 or older
* Within 24 months of initial injury
* experiencing symptoms of photophobia (light sensitivity), increased photophobia since the injury, or no symptoms of photophobia

Exclusion Criteria:

* moderate or severe concussion
* active infection or inflammation that contradicts the use of soft contact lenses
* subjects unable to safely perform insertion and removal of the contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that improved symptoms of light sensitivity with narrow band (tinted) contact lenses | Baseline, 1 week
  Improvement in the Utah Photophobia Symptom Impact Scale version 2 (UPSIS-2) on a scale of 15-60. Anything over 26 is considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Candice I Turner, OD, Principal Investigator — University of Alabama at Birmingham School of Optometry
Locations (1):
- UAB Eye Care, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided